CLINICAL TRIAL: NCT05611229
Title: Real-World Treatment Patterns and Outcomes of Targeted Therapy and Immunotherapy Among BRAF-Positive Melanoma Patients Treated in the Adjuvant Setting and Among BRAF-Positive Metastatic Melanoma Patients With Low Tumor Burden: An Observational Study
Brief Title: Treatment Patterns and Outcomes of Targeted Therapy and Immunotherapy Among BRAF-Positive Melanoma Patients Treated in the Adjuvant Setting and Among BRAF-Positive Metastatic Melanoma Patients With Low Tumor Burden
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS55
Record Dates: First submitted 2022-11-04; First posted 2022-11-09 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Melanoma
Keywords: Adjuvant melanoma,; advanced melanoma,; treatment patterns and outcomes
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Population 1: BRAF+ melanoma patients treated with either TT or IO in the adjuvant setting: Included patients were aged more than or equal to 18 years, were required to have a diagnosis of melanoma (ICD-9 172.x & ICD-10 C43.x or D03.x), pathologic stage III disease, evidence of resection, adjuvant treatment with IO (e.g., nivo or pembro) or TT (e.g., dab+tram) on or after January 1, 2014, and prior to August 30,2020 (data cut-off), and any evidence of a BRAF+ result.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab; Combination Product: Dabrafenib+Trametinib
- Population 2: BRAF+ melanoma patients with LTB treated with TT or IO in the metastatic setting: Included patients were aged more than or equal to 18 years, and were required to have a diagnosis of melanoma (ICD-9 172.x & ICD-10 C43 or D03x), a pathologic stage IV diagnosis, treatment with IO (e.g. ipi, nivo, pembro, ipi+nivo) or TT (dab+tram, vem+cobi, enco+bini) on or after January 1, 2014 and prior to May 31, 2020 (data cut-off), and evidence of a BRAF+ result after therapy initiation. Patients were required to be classified as LTB at the time of stage IV diagnosis. LTB was defined as having normal LDH and <3 metastatic sites at the time of stage IV diagnosis.
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab; Combination Product: Dabrafenib+Trametinib; Combination Product: Ipilimumab+Nivolumab; Combination Product: Vemurafenib+Cobimetinib; Combination Product: Encorafenib+Binimetinib

INTERVENTIONS:
Drug: Nivolumab — Nivolumab
Drug: Pembrolizumab — Pembrolizumab
Combination Product: Dabrafenib+Trametinib — Dabrafenib+Trametinib
Combination Product: Ipilimumab+Nivolumab — Ipilimumab+Nivolumab
  Groups: Population 2: BRAF+ melanoma patients with LTB treated with TT or IO in the metastatic setting
Combination Product: Vemurafenib+Cobimetinib — Vemurafenib+Cobimetinib
  Groups: Population 2: BRAF+ melanoma patients with LTB treated with TT or IO in the metastatic setting
Combination Product: Encorafenib+Binimetinib — Encorafenib+Binimetinib
  Groups: Population 2: BRAF+ melanoma patients with LTB treated with TT or IO in the metastatic setting

SUMMARY:
This was an observational study utilizing electronic health record (EHR)-derived data collected retrospectively during routine care of real-world patients with advanced melanoma from NOBLE (Novartis Braf+ meLanoma patients ObsErvational) dataset.

DETAILED DESCRIPTION:
The NOBLE database was built from the harmonization of two customized oncology specific EHR databases: Flatiron Health Spotlight and Concerto Custom Patient360. BRAF v600 mutated advanced (i.e., stage III or IV) patients treated at oncology practices across the US were identified in these two databases for potential inclusion. Both the Flatiron Health EHR-derived database and the Concerto Patient360 database contain clinical, demographic, treatment, and mortality information for melanoma patients from the time of initial diagnosis until death or the most recent data cut-off, which is August 31, 2020 (for population 1), and May 31, 2020 (for population 2).

For population 1 (patients treated in the adjuvant setting): included patients were aged more than or equal to 18 years, were required to have a diagnosis of melanoma (ICD-9 172.x & ICD-10 C43.x or D03.x), pathologic stage III disease, evidence of resection, adjuvant treatment with Immunotherapy (IO) (e.g., Nivolumab (nivo) or Pembrolizumab (pembro)) or Targeted Therapy (TT) (e.g., Dabrafenib+ Trametinib (dab+tram)) on or after January 1, 2014 and prior to August 30,2020 (data cut-off), and any evidence of a BRAF+ result. Patients were required to have at least 6 months of follow-up after initiation of adjuvant treatment. Patients were followed until the earlier of death, data cut-off, loss of follow-up, or received MM diagnosis. While the first systemic therapy approved for use in the adjuvant melanoma setting occurred in 2015, the study period of interest begins on January 1, 2014, to include any potential off-label use of these therapies as adjuvant therapies.

For population 2 (patients with Low tumor burden (LTB) treated in the metastatic setting): included patients were aged more than or equal to 18 years, and were required to have a diagnosis of melanoma (ICD-9 172.x & ICD-10 C43 or D03x), a pathologic stage IV diagnosis, treatment with IO (e.g. Ipilimumab (ipi), nivo, pembro, ipi+nivo) or TT (dab+tram, Vemurafenib+Cobimetinib, Encorafenib+Binimetinib (vem+cobi, enco+bini) on or after January 1, 2014 and prior to May 31, 2020 (data cut-off), and evidence of a BRAF+ result after therapy initiation. Patients were required to be classified as LTB at the time of stage IV diagnosis. LTB was defined as having normal LDH and <3 metastatic sites at the time of stage IV diagnosis. To align with recent FDA approvals for combination therapies use in the MM setting, the study period of interest began on January 1, 2014. Furthermore, this sampling interval allowed for a maximum of 6 years of follow-up from the start of study period.

ELIGIBILITY:
Inclusion Criteria:

Population 1(patients treated in the adjuvant setting)

* Diagnosis of melanoma (ICD-9 172.x & ICD-10 C43.x or D03.x)
* Pathologic stage III on or after 2011
* Evidence of resection
* Adjuvant treatment with IO (nivo, pembro) or TT (dab+tram) on or after 1/1/2014 and prior to 8/31/2020
* At least 6 months of follow-up time (until death, end of data cut-off, loss-of-follow-up, or progressed to stage IV diagnosis) from the initiation of therapy
* Evidence of a BRAF+ result ≤30 days after therapy initiation in the adjuvant setting
* At least 18 years of age at the time of initiation of treatment
* No documented receipt of a clinical trial treatment for cancer at any time on or after January 1, 2014

Population 2 (patients with LTB treated in the metastatic setting)

* Diagnosis of melanoma (ICD-9 172.x & ICD-10 C43.x or D03.x)
* Pathologic stage IV at initial diagnosis on or after 1/1/2011, or earlier stage disease accompanied by development of a first locoregional recurrence on or after 1/1/2011
* 1L treatment with IO (ipi, nivo, pembro, ipi+nivo) or TT (dab+tram, vemu+cobi, enco+bini) on or after 1/1/2014 and prior to 5/31/2020
* At least 6 months of follow-up time (until death, loss of follow-up, or end of data cut-off) from the initiation of therapy
* Evidence of a BRAF+ result ≤30 days after 1L therapy initiation
* LTB, defined as having <3 involved organ sites and normal LDH test (less than upper limit of normal) at the time of receiving MM diagnosis
* At least 18 years of age at the time of initiation of 1L treatment
* No documented receipt of a clinical trial treatment for cancer at any time on or after 1/1/2014

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world patients with advanced melanoma from NOBLE (Novartis Braf+ meLanoma patients ObsErvational) dataset
Sampling Method: Non-Probability Sample
Enrollment: 1975 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving TT and IO therapy in the first-, and second-line | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020 for population 1 and 01 January 2014 to 31 May 2020 for population 2
  To describe treatment patterns among patients prescribed with TT versus IO in both the populations.
Proportion of patients switching from TT 1L therapy to IO 2L therapy | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020 for population 1 and 01 January 2014 to 31 May 2020 for population 2
  To describe treatment patterns among patients prescribed with TT versus IO in both the populations.
Proportion of patients switching from IO 1L therapy to TT 2L therapy | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020 for population 1 and 01 January 2014 to 31 May 2020 for population 2
  To describe treatment patterns among patients prescribed with TT versus IO in both the populations.

SECONDARY OUTCOMES:
Proportion of patients who discontinued treatment in 1L | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020 for population 1 and 01 January 2014 to 31 May 2020 for population 2
  To evaluate discontinuation of 1L treatment among patients receiving TT or IO.
Reasons for discontinuation of treatment in 1L | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020 for population 1 and 01 January 2014 to 31 May 2020 for population 2
  To evaluate discontinuation of 1L treatment among patients receiving TT or IO.
Time from initiation of 1L therapy to death for any reason | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020 for population 1 and 01 January 2014 to 31 May 2020 for population 2
  To estimate OS from initiation of 1L treatment among patients receiving TT or IO.
Time from initiation of 1L therapy to recurrence (for population 1) | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 30 August 2020)
  To estimate Recurrence Free Survival (RFS) (for population 1) from initiation of 1L treatment among patients receiving TT or IO.
Time from initiation of 1L therapy to progression or death (for population 2) | throughout the study period, approximately 6 years (i.e., 01 January 2014 to 31 May 2020)
  To estimate Progression Free Survival (PFS) (for population 2) from initiation of 1L treatment among patients receiving TT or IO.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CTMT212AUS55 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17991